CLINICAL TRIAL: NCT00879125
Title: Effect of Gastric Bypass on Type 2 Diabetes and/or Dyslipidemia
Brief Title: Effect of Gastric Bypass on Patients With Type 2 Diabetes and/or Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Joan Kaiser, RN, Vanderbilt University
Other Study IDs: 080368
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes
Keywords: Gastric by-pass on patients with T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective review of patients who have undergone bariatric surgery at VUMC and who have type 2 Diabetes and/or dyslipidemia. The investigators have previously found that gastric bypass significantly improves diabetes 6-12 months after surgery. The investigators are interested in looking at the longer term results after surgery.

DETAILED DESCRIPTION:
Review and record changes in the subject's medication. subjects vitals: weight, blood pressure, and fasting blood values, which include:

* HbA1c
* Fasting blood glucose
* Fasting Insulin
* Lipid Panel ( total cholesterol, LDL, HDL and triglycerides) were obtained.

ELIGIBILITY:
Inclusion Criteria:

Patients who have had diabetes and/or dyslipidemia prior to gastric by-pass. -

Exclusion Criteria:Patients who have had type 2 diabetes that was diet controlled at time of surgery; and debilitated patients who are unable to come in for a physical exam.

-

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Type 2 diabetes with a BMI over 35kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 1999-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
glycemic control | one year

SECONDARY OUTCOMES:
Correction of lipid profiles | one year

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States